CLINICAL TRIAL: NCT03488147
Title: The Effect of Esomeprazole Magnesium on Incidence of Dysphagia Following Anterior Cervical Spine Surgery: A Prospective, Randomized, Double Blinded, Placebo-Controlled Study
Brief Title: Whether Proton Pump Inhibitors, Administered Prior to or After Surgery, Can Reduce the Incidence and/or Severity of Difficulty Swallowing Foods and/or Liquids,Following Anterior Cervical Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in Investigational Drug Service policies resulting in the need to change the operational design of the overall protocol.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Andrew Hecht, Assistant Professor, Chief, Spine Surgery, Director, Mount Sinai Spine Center, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 12-1433
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Dysphagia; GERD; Degenerative Joint Disease
Keywords: Esomeprazole Magnesium; Postoperative dysphagia; Gastroesophageal reflux disease; Anterior cervical surgery; Proton pump inhibitor
MeSH Terms: conditions — Deglutition Disorders; Gastroesophageal Reflux; Joint Diseases | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: After consent has been obtained, eligible subjects will be randomized into 1 of 3 different treatment groups designated A, B, and C, using a random number generator.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects assigned to the treatment group 'A' will receive one 20 mg esomeprazole tablet daily starting 1 week prior to the cervical operation and will continue to receive the esomeprazole until the end of the study (12 week follow-up).
  Subjects belonging to the treatment group 'B' will receive one placebo tablet (physically resembling a 20 mg esomeprazole tablet) daily starting one week prior to the cervical operation. Subjects will then receive one 20 mg esomeprazole daily starting immediately after the operation and will continue to receive the esomeprazole until the end of the study.
  Subjects belonging to the treatment group 'C' will receive one placebo tablet (physically resembling a 20 mg esomeprazole tablet) daily starting one week prior to the cervical operation and will continue to receive the placebo tablet until the end of the study (12 week follow-up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Esomeprazole Only (Experimental): Subjects assigned to the treatment group 'A' will receive one 20 mg esomeprazole tablet daily starting 1 week prior to the cervical operation and will continue to receive the esomeprazole until the end of the study
  Interventions: Drug: Esomeprazole
- Esomeprazole and Placebo Oral Tablet (Active Comparator): Subjects belonging to the treatment group 'B' will receive one placebo tablet (physically resembling an esomeprazole tablet 20 mg ) daily starting one week prior to the cervical operation. Subjects will then receive one 20 mg esomeprazole daily starting immediately after the operation and will continue to receive the esomeprazole until the end of the study.
  Interventions: Drug: Esomeprazole; Drug: Placebo Oral Tablet
- Placebo Oral Tablet Only (Placebo Comparator): Subjects belonging to the treatment group 'C' will receive one placebo tablet (physically resembling a 20 mg esomeprazole tablet) daily starting one week prior to the cervical operation and will continue to receive the placebo tablet until the end of the study
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Esomeprazole — 20 mg esomeprazole tablet
  Arms: Esomeprazole Only; Esomeprazole and Placebo Oral Tablet
Drug: Placebo Oral Tablet — resembling esomeprazole tablet
  Arms: Esomeprazole and Placebo Oral Tablet; Placebo Oral Tablet Only

SUMMARY:
The researchers wish to investigate whether proton pump inhibitors, administered prior to or after surgery, can reduce the incidence and/or severity of difficulty swallowing foods and/or liquids,following anterior cervical surgery.

DETAILED DESCRIPTION:
Over half of patients who underwent anterior cervical surgery may experience dysphagia in the month following the operation. Dysphagia, characterized as difficulty swallowing foods and/or liquids, is a debilitating condition that not only reduces the quality of life for our patients but also results in poor nutritional intake, which may lead to delays in healing and recovery after surgery.

Current understanding of dysphagia following cervical surgery is very rudimentary. Many published reports were retrospective studies where the incidence of dysphagia was later found to be greatly underreported. Furthermore, many studies utilized small sample sizes producing varying data regarding the incidence and severity of postoperative dysphagia. Most importantly, a review of the medical literature failed to find any consistently proven recommendations or therapies that can reduce the incidence or severity of postoperative dysphagia.

A recently published study shows that gastroesophageal reflux disease (GERD) is also a common complaint following anterior cervical surgery. The study also shows a positive correlation between the severity of postoperative GERD and severity of postoperative dysphagia. Other studies also showed that patients suffering from GERD-associated dysphagia may be successfully treated with proton pump inhibitors. Based on these studies, along with anecdotal reports, the investigators hypothesize that proton pump inhibitors may reduce the incidence and/or severity of dysphagia following anterior cervical surgery.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* Scheduled to undergo anterior cervical surgery for degenerative joint disease.

Exclusion Criteria:

* Patients undergoing revision procedures, multi-level procedures, or procedures treating conditions other than degenerative joint disease.
* Patients with preoperative dysphagia.
* Patients currently taking any acid suppressing medications (proton pump inhibitors, H2 blockers, antacids, etc).
* Patients who are pregnant or nursing.
* Patients who, due to drug allergies, hypersensitivities/anaphylactic reactions to esomeprazole or contraindications (hypersensitivity to benzimidazoles, osteoporosis), are unable to take esomeprazole.
* Patients unable to attend follow-up visits or answer the dysphagia questionnaires.

Eligibility Criteria:

* Scheduled to undergo anterior cervical surgery for degenerative joint disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Dysphagia questionnaire | 12 weeks post surgery
  The Dysphagia questionnaire is a 2 item questionnaire with full scale from 0 (no swallowing difficulty) to 10 (frequent swallowing difficulty)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Hecht, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York